CLINICAL TRIAL: NCT05860296
Title: An Open-Label, Phase 1b/2a Study of SLC-391, an AXL Inhibitor, in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Testing Experimental Anti-cancer Drug SLC-391 With an Approved Immunotherapy Drug, Pembrolizumab, for Advanced Lung Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy and enrollment challenges
Sponsor: SignalChem Lifesciences Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SLC-391-102; KEYNOTE-C62 (Other: Merck Sharp & Dohme LLC); MK3475-C62 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-04-27; First posted 2023-05-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer Stage IV; Lung Cancer Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Phase 1b Dose Level 1) (Experimental): Dose level 1 dose will be SLC-391 100 mg PO/BID on Days 1-21 of each cycle and Pembrolizumab 200 mg IV on Day 1 of each cycle.
  All dose-escalation decisions and the rationale for progressing to the next cohort will be reviewed by the Safety Review Committee (SRC).
  A subject may continue treatment with SLC-391 and pembrolizumab in 21-day cycles until the treatment discontinuation criteria are met.
  Interventions: Drug: SLC-391; Biological: pembrolizumab
- Dose Escalation (Phase 1b Dose Level 2) (Experimental): Dose level 2 dose will be SLC-391 150 mg PO/BID on Days 1-21 of each cycle and Pembrolizumab 200 mg IV on Day 1 of each cycle.
  All dose-escalation decisions and the rationale for progressing to the next cohort will be reviewed by the Safety Review Committee (SRC).
  Interventions: Drug: SLC-391; Biological: pembrolizumab
- Dose Escalation (Phase 1b Dose Level -1) (Experimental): Dose level -1 dose will be SLC-391 50 mg PO/BID on Days 1-21 of each cycle and Pembrolizumab 200 mg IV on Day 1 of each cycle.
  All dose-escalation decisions and the rationale for progressing to the next cohort will be reviewed by the Safety Review Committee (SRC).
  Interventions: Drug: SLC-391; Biological: pembrolizumab
- ICI-Naïve (Phase 2a) (Experimental): The dose of SLC-391 will be randomized between two dose levels (50 mg and 100 mg PO/BID) as approved by the SRC in combination with Pembrolizumab.
  * Tumors must have PD-L1 expression (TPS ≥1%)
  * No prior systemic treatment (chemotherapy or targeted therapy) and no prior immunotherapy (SOC or investigational) in advanced or metastatic setting
  * Subjects with actionable genomic alterations with approved targeted therapy in first line setting are not allowed
  * Subjects with disease recurrence or progression following neoadjuvant or adjuvant therapy or definitive chemoradiation therapy are eligible.
  * Prior adjuvant, neoadjuvant immunotherapy allowed if completed more than 12 months before documented relapse
  A subject may continue treatment with SLC-391 and pembrolizumab in 21-day cycles until the treatment discontinuation criteria are met.
  Interventions: Drug: SLC-391; Biological: pembrolizumab
- ICI-Resistant (Phase 2a) (Experimental): The dose of SLC-391 will be randomized between two dose levels (50 mg and 100 mg PO/BID) as approved by the SRC in combination with Pembrolizumab.
  * Received at least 2 doses of anti-PD(L)-1 monoclonal antibody (mAb) in an advanced or metastatic setting.
  * Progressive disease documented during treatment or within 12 weeks from the last dose of anti-PD(L)-1 mAb.
  * Maximum of 2 prior lines of cancer therapy in an advanced or metastatic setting including an anti-PD(L)-1 mAb administered either as monotherapy or in combination with other therapies.
  * Subjects who received a targeted therapy for an actionable genomic alteration can participate with documented disease progression or if unable to tolerate the targeted therapy. Only these subjects are allowed to receive up to a maximum of 3 prior lines of cancer therapy in an advanced or metastatic setting.
  A subject may continue treatment with SLC-391 and pembrolizumab in 21-day cycles until the treatment discontinuation criteria are met.
  Interventions: Drug: SLC-391; Biological: pembrolizumab

INTERVENTIONS:
Drug: SLC-391 — SLC-391 is an AXL inhibitor
Biological: pembrolizumab — Immunotherapy
  Other Names: KEYTRUDA®

SUMMARY:
SLC-391 is a novel, potent and specific small molecule inhibitor of receptor tyrosine kinase AXL with desirable potency and pharmaceutical properties.

The study is being done to evaluate the safety and pharmacokinetic (PK) profile of SLC-391 in combination with pembrolizumab in participants with non-small cell lung cancer (NSCLC).

Each treatment cycle lasts 21 days. Participants will swallow SLC-391 pills two times every day. Participants will get pembrolizumab intravenously (IV) from the study site staff on the first day of every cycle.

This study has 2 parts. The first part will determine the recommended dose of SLC-391 in combination with pembrolizumab. The second part wants to find out if the combination of SLC-391 and pembrolizumab can help stop NSCLC tumours from growing or spreading.

ELIGIBILITY:
Inclusion Criteria:

* The subject provides written informed consent.
* Adults ≥ 18 years of age on day of signing informed consent.
* Disease must be measurable per RECIST 1.1, as assessed by the Site(s) Investigator/radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in these lesions.
* Subject has histologically or cytologically documented, locally advanced (Stage IIIB or IIIC) disease (not candidate for surgical resection, local therapies with curative intent, or definitive chemoradiation) or the subject has metastatic NSCLC (Stage IV). Staging will be based on the American Joint Committee on Cancer, Eighth Edition. Subjects with adenocarcinoma, large cell carcinoma, undifferentiated carcinoma, squamous carcinoma, or mixed histology are eligible. Subjects with a small cell component are not eligible.
* Phase 1b Subjects additional eligibility criteria:

  1. Subjects must have received a minimum of one prior systemic treatment for advanced unresectable or metastatic NSCLC and progressed following prior SOC.
  2. Maximum of up to 4 prior lines of therapy in an advanced or metastatic setting is allowed.
  3. Subjects who had disease recurrence or progression following neoadjuvant or adjuvant therapy or definitive chemoradiation therapy are eligible.
  4. Subjects who received treatment with an approved/available targeted therapy for an actionable genomic alteration (including but not limited to EGFR, ALK, ROS1, KRAS, etc.) can participate if they have documented disease progression or were unable to tolerate the approved targeted therapy.

Phase 1b Notes:

* Targeted therapy for advanced setting is counted as a prior line of therapy.
* Prior use of a PD(L)-1, anti-CTLA-4 (Cytotoxic T-lymphocyte associated protein 4) antibody, or any other antibody or drug that specifically targets immune checkpoint pathway is allowed and is counted as a prior line of therapy.
* Neoadjuvant and adjuvant therapies initiated < 12 months prior to the first dose of study drug(s) will be counted as one prior line of therapy for advanced setting.
* Neoadjuvant and adjuvant therapies initiated ≥ 12 months prior to the first dose of study drug(s) are not counted as prior lines of therapy.
* Maintenance therapy is not counted as a prior line of therapy.
* Phase 2a Subjects additional eligibility criteria:

Cohort 1:

1. Tumors must have PD-L1 expression (TPS ≥ 1% as determined by SOC).
2. Subjects are eligible to participate if they did not receive any prior therapy (SOC or investigational) or prior immunotherapy of any kind for advanced or metastatic disease. See Exclusion Criteria 1.0.
3. Subjects with disease recurrence or progression following neoadjuvant or adjuvant therapy or definitive chemoradiation therapy are eligible.
4. Prior adjuvant or neoadjuvant immunotherapy is allowed if completed more than 12 months before documented relapse.

Cohort 2:

1. Subjects should have received at least 2 doses of an approved anti PD(L) 1 monoclonal antibody (mAb) in an advanced or metastatic setting.
2. Progressive disease should be documented during treatment or within 12 weeks from the last dose of anti-PD(L)-1 mAb.
3. Up to a maximum of 2 prior lines of approved cancer therapy in an advanced or metastatic setting, including an anti-PD(L)-1 mAb administered either as monotherapy or in combination with other therapies, is allowed.
4. Subjects who received treatment with an approved/available targeted therapy for an actionable genomic alteration (including but not limited to EGFR, ALK, ROS1, KRAS, etc.) can participate if they have documented disease progression or were unable to tolerate the approved targeted therapy. Only these subjects are allowed to receive up to a maximum of 3 prior lines of cancer therapy in an advanced or metastatic setting.
5. Subjects with disease recurrence or progression following neoadjuvant or adjuvant therapy or definitive chemoradiation therapy are eligible.

Cohort 2 Notes:

* Targeted therapy for advanced setting is counted as a prior line of therapy.
* Maintenance therapy is not counted as a prior line of therapy.
* Neoadjuvant and adjuvant therapies initiated < 12 months prior to first dose of study drug(s) will be counted as one prior line of therapy for advanced setting.
* Neoadjuvant and adjuvant therapies initiated ≥ 12 months prior to first dose of study drug(s) are not counted as prior lines of therapy.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 3 months.
* An archival tumor tissue sample or newly obtained biopsy of a tumor lesion not previously irradiated must exist to participate in the study (Mandatory in Phase 2a but subjects in Phase 1b may be enrolled in the absence of a tumor tissue sample). Only core needle and/or excisional biopsy samples, from archival or fresh tissue, will be accepted in this study.
* Adequate organ function as defined below must be met for subjects to participate in the study. Clinical laboratory specimens must be collected within 10 days prior to first dose of study drug(s):

  1. Absolute neutrophil count (ANC) ≥ 1500/µL or ≥ 1.5 × 109/L (in the absence of growth factor support).
  2. Platelets ≥ 100,000/µL or 100 × 109/L (in the absence of transfusion or growth factor support).
  3. Hemoglobin ≥ 9 g/dL or ≥ 90 g/L (in the absence of transfusion). Note: Criteria must be met without packed red blood cell transfusion within the prior 2 weeks. Subjects can be on stable dose of erythropoietin (≥ approximately 3 months).
  4. Creatinine Clearance (CCr) ≥ 50 mL/minute using the Cockcroft and Gault formula.

     Note: The Cockcroft and Gault formula (1973): CCr = ([{140 - age} × weight]/[72 × SCr]) × 0.85 (if female); where CCr = mL/minute; age = years; weight = kg; SCr (serum creatinine) = mg/dL.
  5. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (unless a diagnosis of Gilbert's syndrome in which case ≤ 3 × ULN) OR direct bilirubin ≤ 1 × ULN for participants with total bilirubin >1.5 × ULN.
  6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5× ULN for subjects with liver metastases).
  7. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN; if the subject is receiving anticoagulant therapy PT or INR should be within the therapeutic range of the intended use of anticoagulants.
  8. Activated partial thromboplastin time/partial thromboplastin time (aPTT/PTT) ≤ 1.5 × ULN; if the subject is receiving anticoagulant therapy PTT should be within the therapeutic range of intended use of anticoagulants.

Note: Low molecular weight heparin, warfarin (INR monitoring required), direct oral anticoagulants, and drugs in the anticoagulant class (e.g., Lovenox [enoxaparin]) administered for deep vein thrombosis are permitted.

* Women who are not of childbearing potential must be documented and will not be tested for pregnancy or required to utilize contraception if they meet one or more of the following definitions of non-childbearing potential:

  1. Amenorrheic for > 2 years without a hysterectomy and oophorectomy, and a follicle stimulating hormone (FSH) value in the postmenopausal range upon screening evaluation.
  2. Post-hysterectomy, bilateral oophorectomy, or tubal ligation. Tubal ligation should be confirmed with medical records of the actual procedure.
* 12. Women of childbearing potential (WOCBP) must have a negative pregnancy test (serum) within 72 hours prior to first dose of study drug(s) and meet the following criteria throughout the study, starting with the screening visit through 120 days after the last dose of study drug(s) (or 30 days if new cancer therapy is initiated):

  1. Agrees to follow contraceptive guidance throughout the study as per protocol.
  2. Willing to use 2 highly effective birth control methods throughout the study. The 2 birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Refer to Appendix 4 for complete list of acceptable birth control methods.
  3. Refrain from egg donation. Note: If there is any question that a subject will not reliably comply with the requirements for contraception, that subject should not be enrolled.
* Male subjects must agree to use an acceptable method of contraception and refrain from sperm donation throughout the study: from screening, during the treatment period, and for at least 120 days after the last dose of study drug(s) (or 30 days if new cancer therapy is initiated).
* Willing and able to participate in blood sampling and all other required study procedures.

Exclusion Criteria:

* Phase 2a - Cohort 1 (only) exclusion criteria:

  1. Subjects have tumors that have actionable genomic alterations with approved targeted therapy in first line setting are not eligible to participate.
  2. Subjects are not eligible if they received any prior therapy (SOC or investigational) for advanced or metastatic disease including chemotherapy, targeted therapy, or immunotherapy of any kind such as the following: pembrolizumab, an anti-PD(L)-1 or anti-programmed death ligand 2 (PD-L2) agent, or an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA4, OX40 (Tumor necrosis factor receptor superfamily, member 4), CD137(Tumor necrosis factor receptor superfamily member 9)).
* Undergone prior treatment with a known AXL inhibitor such as bemcentinib (see Section 8.2.2 for full list of AXL inhibitors).
* Received prior systemic anticancer therapy within 5 half-lives or 3 weeks, whichever is shorter, prior to starting the first dose of study drug(s). Examples of prior systemic anticancer therapy includes cytotoxic agents, targeted therapy such as small molecules, mAbs and hormonal therapy etc..
* Received immunotherapies [including but not limited to PD(L)-1 inhibitors, etc.] within 4 weeks prior to starting the first dose of study drug(s).
* Received prior radiotherapy within 2 weeks of the first dose of study drug(s) or had a history of radiation pneumonitis.

Note: Subjects must have recovered from all radiation-related toxicities and not require corticosteroids. A 1 week washout is permitted following palliative radiation (≤ 2 weeks of radiotherapy) for non-central nervous system (CNS) disease.

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study drug(s).

Note: Subjects who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent, follow-up is primarily non-invasive, and the subject can comply with protocol requirements.

* Has not recovered to ≤ Grade 1 or to baseline from prior cancer therapy toxicity.

Note: Subject with ≤ Grade 2 neuropathy may be an exception to this criterion and may qualify for the study after discussion with Sponsor. Subjects with endocrine-related AEs ≤ Grade 2 requiring treatment or hormone replacement may be eligible after discussion with Sponsor.

Note: Toxic effects also include laboratory results that have not resolved to ≤ Grade 1. Subjects with ≤ Grade 2 alopecia are an exception to this criterion.

* Has not adequately recovered from major surgery and/or complications from the procedure prior to the first dose of study drug(s).
* Pulmonary hemorrhage or hemoptysis > 2.5 mL blood within 6 weeks of screening (or within 2 weeks if the source of bleeding is treated).
* Received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug(s). Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guerin, and typhoid vaccine. Seasonal influenza vaccines are generally killed virus vaccines and are permitted; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live-attenuated vaccines and are not allowed.

Note: The administration of killed vaccines, mRNA vaccines, and DNA vaccines is allowed.

* Has an active diagnosis of immunodeficiency or is receiving systemic steroid therapy (exceeding 10 mg daily of prednisone equivalent) or has received any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug(s).
* Has active autoimmune disease which required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

Note: Hormone therapy (e.g., thyroxine, insulin, or corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

* Known additional malignancy that is progressing or has required active treatment within the past 2 years.

Note: Subjects with curatively treated basal or squamous cell carcinoma of the skin (non-melanoma skin cancer), cervical or vaginal intra-epithelial neoplasia, non-invasive breast cancer in situ, or localized prostate cancer with a prostate-specific antigen level of < 4 ng/mL (µg/L) at screening are not excluded. Subjects with other curatively treated malignancies who have had a > 2-year disease-free interval and whose natural history or treatment does not have the potential to interfere with investigational agents (e.g., hormone maintenance) may be enrolled after approval by the Medical Monitor/Sponsor.

* Known active CNS metastases and/or carcinomatous meningitis. Subjects with adequately treated brain metastases may participate provided they meet the following criteria:

  1. Are radiologically stable (no progression) for at least 4 weeks as documented by screening computed tomography (CT) or magnetic resonance imaging (MRI) scan.
  2. Clinically stable.
  3. No evidence of new or enlarging brain metastases. Does not require steroids for at least 14 days before starting first dose of study drug(s) (anticonvulsants at a stable dose are allowed). Low dose steroids equivalent of prednisone ≤ 10 mg orally once a day is allowed.
  4. No history of intracranial or spinal cord hemorrhage.
  5. No evidence of significant vasogenic edema.
* Severe hypersensitivity (≥ Grade 3) to pembrolizumab or SLC-391 and/or any excipients.
* A history of non-infectious pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* A known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies). No HIV testing is required unless mandated by the local health authority.
* Known history of Hepatitis B (Anti-HBc and HBsAg reactive) or known active Hepatitis C virus (RNA, qualitative) infection.

Note: No testing for Hepatitis B or C is required unless mandated by a local health authority.

* A history or current evidence of any severe acute or chronic medical or psychiatric condition that requires treatment, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject, in the opinion of the Principal Investigator (PI; also referred to as Investigator). Examples include, but are not limited to, active uncontrolled infection (including tuberculosis [TB]) requiring systemic therapy, transfusion dependent anemia, recent (within 90 days) stroke or myocardial infarction, unstable angina, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, symptomatic congestive heart failure (New York Heart Association class ≥ III/IV), and recent severe Coronavirus disease 2019 (COVID-19).

Note: TB testing is required for subjects recently exposed to persons with active TB or who have traveled recently to areas where TB is endemic.

* Systolic blood pressure (BP) ≥ 160 mmHg or diastolic BP ≥100 mmHg.
* Has a corrected QT interval by Fridericia (QTcF) ≥ 470 msec. Note: Apply the Fridericia QT correction to calculate QTcF using the following formula: QTcF = QT/RR1/3 where QT = the time between the start of the QRS complex and the end of the T wave and RR = the time between the start of one QRS complex and the start of the next QRS complex.

Note: If a subject has a prolonged QT interval and the prolongation is deemed to be due to a pacemaker as deemed by the Investigator (i.e., the subject otherwise has no cardiac abnormalities), the subject may be eligible to participate in the study following discussion with the Sponsor.

* History or presence of sustained or symptomatic bradycardia (≤ 55 bpm), left bundle branch block, ventricular arrhythmia excluding premature ventricular contractions, or uncontrolled ventricular arrhythmia. Subjects with a supraventricular arrhythmia requiring medical treatment and a normal ventricular rate are eligible.
* Psychological, familial, sociological, or geographical conditions including known psychiatric or substance abuse disorder that could interfere with the subject's ability to provide informed consent, comply with the protocol, or interfere with the interpretation of the study results.
* Inability to swallow oral medication and/or the presence of active gastrointestinal (GI) disease and/or other GI conditions, including bowel resection, that is expected to interfere significantly with the absorption, distribution, metabolism, or excretion of oral SLC-391 therapy.
* Received radiation therapy to the lung that is > 30 Gy within 6 months of the first dose of study drug(s).
* Had an allogenic tissue, marrow, or solid organ transplant.
* Females who are pregnant or nursing. Note: SLC reserves the right to deny any subject enrollment based upon potential safety concern(s) or factors that could confound the study results.

Note: The Investigator or licensed, medically qualified Sub-Investigator must review and confirm eligibility prior to the first dose of study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Determine doses of SLC-391 in combination with pembrolizumab for further evaluation in Phase 2a. | DLTs will be evaluated during the during the first 21 days of treatment Cycle 1 in the Phase 1b portion of the study.
  After a minimum of 3 evaluable subjects have completed the 21-day DLT (Dose Limiting Toxicity) evaluation period, SRC will review all available safety, efficacy, PK, and pharmacodynamic data and determine whether to expand the current dose level or escalate or de-escalate.
  A subject is considered "evaluable" for dose-decisions during Phase 1b if the subject has completed the 21-day DLT evaluation period and has received at least 75% of the planned dose of study drug during the DLT evaluation period, or the subject has experienced a DLT. The number of subjects experiencing a DLT will inform the SRC's decision on whether to expand, escalate or de-escalate.
  AEs are defined using NCI-CTCAE v5.0 and DLTs include events ≥ Grade 3 in severity with some exceptions.
Phase 1b: Number of Participants with Adverse Events (AEs) as assessed by CTCAE V5.0 | From first dose through 90-days following cessation of SLC-391 and pembrolizumab
  To assess AEs as criteria of safety of oral SLC-391 in combination with pembrolizumab
Phase 2a: Antitumor activity of SLC-391 (objective response rate [ORR]) in combination with pembrolizumab, using RECIST version 1.1 | From date of baseline tumor assessment to the date of first documented CR or PR, assessed up to 24 months.
  Proportion of subjects who have achieved complete response (CR) or partial response (PR), evaluated using RECIST 1.1 for tumor assessment.
Phase 2a: Number of Participants with Adverse Events (AEs) as assessed by CTCAE V5.0 | From first dose through 90-days following cessation of SLC-391 and pembrolizumab
  To assess AEs as criteria of safety of oral SLC-391 in combination with pembrolizumab(PR), evaluated using RECIST 1.1 for tumor assessment.

SECONDARY OUTCOMES:
Phase 2a: Optimal Biological Dose (OBD) of SLC-391 in combination with pembrolizumab. | Up to 24 months
  Optimal Biological Dose
Phase 1b and Phase 2a: Number of Participants with Adverse Events (AEs) as assessed by CTCAE V5.0 | From first dose through 90-days following cessation of SLC-391 and pembrolizumab
  To assess AEs as criteria of safety of oral SLC-391 in combination with pembrolizumab
Phase 1b and Phase 2a: Plasma levels of SLC-391 when administered in combination with pembrolizumab | On Day 1 of Cycles 1,2,4,6,8,10,12 (each cycle is 21 days) and the date of first objective response by RECIST 1.1, assessed up to 24 months.
  Pharmacokinetics of blood sample (plasma) levels of SLC-391 will be analyzed using validated high-performance liquid chromatography with tandem quadrupole mass spectrometry detection
Phase 1b: ORR of participants treated with SLC-391 in combination with pembrolizumab | Up to 24 months
  ORR by RECIST (RECIST) as assessed by investigators. Defined as the proportion of subjects who have achieved complete response (CR) or partial response (PR), evaluated using RECIST 1.1 based on Investigator assessment.
Phase 1b and Phase 2a: Disease control rate (DCR) of participants treated with SLC-391 in combination with pembrolizumab | Up to 24 months
  Disease control rate (DCR) by RECIST 1.1 as assessed by investigators. Defined as as the percentage of subjects achieving CR, PR, or SD (Stable disease) as assessed by the Investigator per RECIST 1.1.
Phase 1b and Phase 2a:Time-to-response (TTR) of participants treated with SLC-391 in combination with pembrolizumab | From the date of first dose of study drug(s) to the date of first objective response by RECIST 1.1, assessed up to 24 months.
  Time-to-response (TTR) by RECIST 1.1 as assessed by investigators.
Phase 1b and Phase 2a: Duration of response (DoR) of participants treated with SLC-391 in combination with pembrolizumab | From date of first objective response to the date of first objective evidence of disease progression or death by RECIST 1.1, assessed up to 24 months.
  Duration of response (DoR) by RECIST 1.1 as assessed by investigators
Phase 1b and Phase 2a: Progression-free survival (PFS) of participants treated with SLC-391 in combination with pembrolizumab | From the date of first dose of study drug(s) to the date of first objective evidence of disease progression or death from any cause, whichever is earlier, assessed up to 24 months.
  Progression-free survival (PFS) by RECIST 1.1 as assessed by investigators
Phase 1b and Phase 2a: Time-to-progression (TTP) of participants treated with SLC-391 in combination with pembrolizumab | From the date of the first dose of study drug(s) to the date of first objective evidence of disease progression by RECIST 1.1, assessed up to 24 months.
  Time-to-progression (TTP) by RECIST 1.1 as assessed by investigators
Phase 1b and Phase 2a: Overall Survival (OS) of participants treated with SLC-391 in combination with pembrolizumab | From the date of first dose to the date of death by any cause, assessed up to 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Zaihui Zhang, PhD, Study Director — SignalChem LifeSciences
Locations (12):
- United States (6):
  - Community Health Network, Indianapolis, Indiana
  - Horizon Verdi Oncology, Lafayette, Indiana
  - Karmanos Cancer Center, Detroit, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Morrison D, Lu L, Singh M, Yan J, Leighl N, Laurie SA, Hotte S. First-in-Human Phase I Clinical Trial of SLC-391, a Novel and Selective AXL Inhibitor, in Patients with Advanced Solid Tumours. Pharmaceuticals (Basel). 2025 Dec 17;18(12):1898. doi: 10.3390/ph18121898. PMID 41471387